CLINICAL TRIAL: NCT02709109
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled, Incomplete Block, Crossover Study to Evaluate the Safety and Efficacy of VX-371 in Subjects Aged 12 Years or Older With Cystic Fibrosis, Homozygous for the F508del-CFTR Mutation, and Being Treated With Orkambi
Brief Title: A Study to Evaluate the Safety and Efficacy of VX-371 in Subjects With Cystic Fibrosis Who Are Homozygous for the F508del-CFTR Mutation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Parion Sciences (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: VX15-371-101; 2015-004841-13 (EudraCT Number)
Record Dates: First submitted 2016-02-29; First posted 2016-03-15 (Estimated); Results first posted 2021-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic; lumacaftor, ivacaftor drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence 1: VX-371 + Hypertonic Saline (HS), then HS (Experimental): Participants received 85 microgram (mcg) VX-371 diluted in 3 milliliter (mL) 4.2 percent (%) HS through oral nebulized inhalation twice daily for 28 days (Day 1 to Day 28) in treatment period 1 followed by a 28 days washout period (Day 29 to Day 56) and then received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (Day 57 to Day 84) in treatment period 2. Participants also received a stable dose of 2 tablets of Orkambi (lumacaftor 400 milligram (mg)/ivacaftor 250 mg) orally every 12 hours with fat-containing food throughout the study as part of their cystic fibrosis (CF) standard of care.
  Interventions: Drug: VX-371 + HS; Drug: Hypertonic saline; Drug: Orkambi
- Sequence 2: HS, then VX-371 + HS (Experimental): Participants received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (Day 1 to Day 28) in treatment period 1 followed by a 28 days washout period (Day 29 to Day 56) and then received 85 mcg VX-371 diluted in 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (Day 57 to Day 84) in treatment period 2. Participants also received a stable dose of 2 tablets of Orkambi (lumacaftor 400 mg/ivacaftor 250 mg) orally every 12 hours with fat-containing food throughout the study as part of their CF standard of care.
  Interventions: Drug: VX-371 + HS; Drug: Hypertonic saline; Drug: Orkambi
- Sequence 3: VX-371 + Placebo, then Placebo (Experimental): Participants received 85 mcg VX-371 diluted in 3 mL 0.17% Saline (placebo) through oral nebulized inhalation twice daily for 28 days (Day 1 to Day 28) in treatment period 1 followed by a 28 days washout period (Day 29 to Day 56) and then received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (Day 57 to Day 84) in treatment period 2. Participants also received a stable dose of 2 tablets of Orkambi (lumacaftor 400 mg/ivacaftor 250 mg) orally every 12 hours with fat-containing food throughout the study as part of their CF standard of care.
  Interventions: Drug: Placebo; Drug: Orkambi; Drug: VX-371
- Sequence 4: Placebo, then VX-371 + Placebo (Experimental): Participants received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (Day 1 to Day 28) in treatment period 1 followed by a 28 days washout period (Day 29 to Day 56) and then received 85 mcg VX-371 diluted in 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days (Day 57 to Day 84) in treatment period 2. Participants also received a stable dose of 2 tablets of Orkambi (lumacaftor 400 mg/ivacaftor 250 mg) orally every 12 hours with fat-containing food throughout the study as part of their CF standard of care.
  Interventions: Drug: Placebo; Drug: Orkambi; Drug: VX-371

INTERVENTIONS:
Drug: VX-371 + HS
  Arms: Sequence 1: VX-371 + Hypertonic Saline (HS), then HS; Sequence 2: HS, then VX-371 + HS
Drug: Hypertonic saline
  Arms: Sequence 1: VX-371 + Hypertonic Saline (HS), then HS; Sequence 2: HS, then VX-371 + HS
Drug: Placebo
  Arms: Sequence 3: VX-371 + Placebo, then Placebo; Sequence 4: Placebo, then VX-371 + Placebo
Drug: Orkambi
  Other Names: lumacaftor/ivacaftor
Drug: VX-371
  Arms: Sequence 3: VX-371 + Placebo, then Placebo; Sequence 4: Placebo, then VX-371 + Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of treatment with VX-371 in hypertonic saline compared to hypertonic saline alone in subjects with cystic fibrosis (CF) who are ≥12 years of age, homozygous for the F508del-cystic fibrosis transmembrane conductance regulator (CFTR) mutation, and being treated with Orkambi

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to use the delivery device as directed by the study manual.
* Confirmed diagnosis of CF, defined as a sweat chloride value ≥60 mmol/L by quantitative pilocarpine iontophoresis.
* Homozygous for the F508del CFTR mutation. If the CFTR screening genotype result is not received before randomization, a previous CFTR genotype lab report may be used to establish eligibility.
* Percent predicted forced expiratory volume at one second (FEV1) of ≥40 to <90 percentage points adjusted for age, sex, and height according to the Global Lung Initiative (GLI) at the Screening Visit.
* Willing to discontinue physician-prescribed saline use.
* Female subjects of childbearing potential with a negative serum pregnancy test at the Screening Visit.

Exclusion Criteria:

* History of any comorbidity, which in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject.
* Any clinically significant laboratory abnormalities at the Screening Visit that would interfere with the study assessments or pose an undue risk for the subject.
* An acute upper or lower respiratory infection, pulmonary exacerbation, or changes in therapy (including antibiotics) for pulmonary disease within 28 days before Day 1 (first dose of study drug).
* A 12 lead ECG demonstrating QTcF >450 msec at the Screening Visit.
* History of solid organ or hematological transplantation.
* Used diuretics or renin-angiotensin aldosterone system antihypertensive drugs in the 28 days prior to Screening or an anticipated need for any of these medications during the study.
* Ongoing or prior participation in an investigational drug study within 30 days of the Screening Visit.
* Inability to withhold short-acting, long-acting, or once-daily, long-acting bronchodilator use for 4, 12, or 24 hours prior to clinic visit, respectively.
* History of significant intolerance to inhaled saline, or intolerance to the single dose of saline at Screening
* Known hypersensitivity or history of intolerance to Orkambi.
* Pregnant and nursing females.
* Subjects who have participated in Parion Sciences Study NCT02343445.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2016-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Church, MD, Study Chair — Parion Sciences
Locations (40):
- United States (30):
  - Little Rock, Arkansas
  - Oakland, California
  - Gainesville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Chicago, Illinois
  - Glenview, Illinois
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Grand Rapids, Michigan
  - Minneapolis, Minnesota
  - Jackson, Mississippi
  - Lebanon, New Hampshire
  - Albuquerque, New Mexico
  - Albany, New York
  - Hawthorne, New York
  - Syracuse, New York
  - Charlotte, North Carolina
  - Cleveland, Ohio
  - Pittsburgh, Pennsylvania
  - Austin, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- France (4):
  - Bron
  - Pierre-Bénite
  - Roscoff
  - Strasbourg
- Dublin, Ireland
- United Kingdom (5):
  - Birmingham
  - Bristol
  - London
  - Manchester
  - Southampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 147 participants entered in this study, 5 participants discontinued from the study before the randomization. Of which 142 participants were randomized to receive 1 of the 4 treatment sequences: 1) VX-371 + hypertonic saline (HS), Then HS; 2) HS, Then VX-371 + HS; 3) VX-371 + Placebo, Then Placebo; 4) Placebo, Then VX-371 + Placebo.
Groups:
- Sequence 1: VX-371 + HS, Then HS: Participants received 85 microgram (mcg) VX-371 diluted in 3 milliliter (mL) 4.2 percent (%) HS through oral nebulized inhalation twice daily for 28 days (Day 1 to Day 28) in treatment period 1 followed by a 28 days washout period (Day 29 to Day 56) and then received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (Day 57 to Day 84) in treatment period 2. Participants also received a stable dose of 2 tablets of Orkambi (lumacaftor 400 milligram (mg)/ivacaftor 250 mg) orally every 12 hours with fat-containing food throughout the study as part of their cystic fibrosis (CF) standard of care.
Period: Treatment Period 1 (28 Days)
Arm/Group | Sequence 1: VX-371 + HS, Then HS | Sequence 2: HS, Then VX-371 + HS | Sequence 3: VX-371 + Placebo, Then Placebo | Sequence 4: Placebo, Then VX-371 + Placebo
Started | 49 | 47 | 22 | 24
Completed | 45 | 42 | 21 | 24
Not Completed | 4 | 5 | 1 | 0
Not completed — Adverse Event | 3 | 3 | 1 | 0
Not completed — Participant refused further dosing | 0 | 2 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0
Period: Washout Period (28 Days)
Arm/Group | Sequence 1: VX-371 + HS, Then HS | Sequence 2: HS, Then VX-371 + HS | Sequence 3: VX-371 + Placebo, Then Placebo | Sequence 4: Placebo, Then VX-371 + Placebo
Started | 45 | 42 | 21 | 24
Completed | 43 | 40 | 18 | 24
Not Completed | 2 | 2 | 3 | 0
Not completed — Other | 2 | 2 | 3 | 0
Period: Treatment Period 2 (28 Days)
Arm/Group | Sequence 1: VX-371 + HS, Then HS | Sequence 2: HS, Then VX-371 + HS | Sequence 3: VX-371 + Placebo, Then Placebo | Sequence 4: Placebo, Then VX-371 + Placebo
Started | 43 | 40 | 18 | 24
Completed | 41 | 36 | 15 | 24
Not Completed | 2 | 4 | 3 | 0
Not completed — Adverse Event | 2 | 3 | 0 | 0
Not completed — Other non-compliance | 0 | 1 | 1 | 0
Not completed — Requires prohibited medication | 0 | 0 | 1 | 0
Not completed — Other | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all randomized participants who carried the intended homozygous F508del-CFTR mutation and received at least 1 dose of inhaled study drug.
Groups:
- Sequence 1: VX-371 + HS, Then HS: Participants received 85 mcg VX-371 diluted in 3 milliliter (mL) 4.2% HS through oral nebulized inhalation twice daily for 28 days (Day 1 to Day 28) in treatment period 1 followed by a 28 days washout period (Day 29 to Day 56) and then received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days (Day 57 to Day 84) in treatment period 2. Participants also received a stable dose of 2 tablets of Orkambi (lumacaftor 400 mg/ivacaftor 250 mg) orally every 12 hours with fat-containing food throughout the study as part of their CF standard of care.
- Total: Total of all reporting groups
Arm/Group | Sequence 1: VX-371 + HS, Then HS | Sequence 2: HS, Then VX-371 + HS | Sequence 3: VX-371 + Placebo, Then Placebo | Sequence 4: Placebo, Then VX-371 + Placebo | Total
Number analyzed (Participants) | 49 | 47 | 22 | 24 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.6 (9.07) | 22.3 (8.75) | 26.0 (10.95) | 22.1 (7.80) | 23.3 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 16 | 7 | 11 | 55
  Male | 28 | 31 | 15 | 13 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 45 | 22 | 23 | 139
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 49 | 45 | 22 | 23 | 139
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. AEs included abnormal clinically significant findings for spirometry, clinical laboratory parameters, standard 12-lead electrocardiograms (ECGs), vital signs and ophthalmologic examinations. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 112 days (up to 28 days after last dose) that were absent before treatment or that worsened relative to pretreatment state. TEAEs included both serious and non-serious TEAEs.
Time Frame: Baseline (Day 1) up to 28 days post last administration of study drug (up to 112 days)
Population: Safety set included all participants who received at least 1 dose of inhaled study drug.
Measure: Count of Participants; unit: Participants
Groups:
- VX-371 + Hypertonic Saline: Participants received 85 mcg VX-371 diluted in 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
- Hypertonic Saline: Participants received 3 mL 4.2% HS through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
- VX-371 + Placebo: Participants received 85 mcg VX-371 diluted in 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
- Placebo: Participants received 3 mL 0.17% saline (placebo) through oral nebulized inhalation twice daily for 28 days in either treatment period 1 or 2.
Arm/Group | VX-371 + Hypertonic Saline | Hypertonic Saline | VX-371 + Placebo | Placebo
Number analyzed (Participants) | 89 | 90 | 46 | 42
Participants
  Participants With TEAEs | 65 | 66 | 32 | 28
  Participants With Serious TEAEs | 8 | 4 | 6 | 3

2. Primary Outcome: Absolute Change From Study Baseline in Percent Predicted Forced Expiratory Volume in 1 Second (ppFEV1) at Day 28
Description: FEV1 is the volume of air that can forcibly be blown out in one second, after full inspiration. Study Baseline was defined as the most recent non-missing measurement before the first dose of inhaled study drug in the study. Day 28 measurements after treatment discontinuation from the treatment period in which discontinuation occurred were included in the analysis.
Time Frame: Study baseline, Day 28
Population: The full analysis set (FAS) included all randomized participants who carried the intended homozygous F508del-cystic fibrosis transmembrane conductance regulator (CFTR) mutation and received at least 1 dose of inhaled study drug. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: percentage points
Arm/Group | VX-371 + Hypertonic Saline | Hypertonic Saline | VX-371 + Placebo | Placebo
Number analyzed (Participants) | 79 | 77 | 43 | 38
percentage points | 0.1 (0.8) | -0.1 (0.8) | -0.8 (1.1) | 0.8 (1.1)
Statistical Analysis 1: Comparison: VX-371 + Hypertonic Saline vs Hypertonic Saline; Test type: Superiority; p = 0.8173, Mixed-effects Model for Repeated Measure; Least Square (LS) mean difference = 0.2, 95% CI 2-sided [-1.4 to 1.8]
Statistical Analysis 2: Comparison: Hypertonic Saline vs VX-371 + Placebo; Test type: Superiority; p = 0.5903, Mixed-effects Model for Repeated Measure; LS mean difference = -0.7, 95% CI 2-sided [-3.3 to 1.9]
Statistical Analysis 3: Comparison: VX-371 + Hypertonic Saline vs Placebo; Test type: Superiority; p = 0.5917, Mixed-effects Model for Repeated Measure; LS mean difference = -0.7, 95% CI 2-sided [-3.4 to 1.9]
Statistical Analysis 4: Comparison: Hypertonic Saline vs Placebo; Test type: Superiority; p = 0.5021, Mixed-effects Model for Repeated Measure; LS mean difference = -0.9, 95% CI 2-sided [-3.6 to 1.8]
Statistical Analysis 5: Comparison: VX-371 + Placebo vs Placebo; Test type: Superiority; p = 0.1382, Mixed-effects Model for Repeated Measure; LS mean difference = -1.6, 95% CI 2-sided [-3.8 to 0.5]
Statistical Analysis 6: Comparison: VX-371 + Hypertonic Saline vs VX-371 + Placebo; Test type: Superiority; p = 0.4962, Mixed-effects Model for Repeated Measure; LS mean difference = 0.9, 95% CI 2-sided [-1.7 to 3.5]

3. Secondary Outcome: Plasma Concentrations of VX-371
Time Frame: Pre-dose (90 minutes prior inhaled study drug administration) and 60 minutes post-dose on Days 1, 14 and 28 within treatment period 1 and 2
Population: The Pharmacokinetic (PK) analysis set included all participants who received at least 1 dose of VX-371. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: Picograms per milliliter (pg/mL)
Arm/Group | VX-371 + Hypertonic Saline | VX-371 + Placebo
Number analyzed (Participants) | 89 | 45
Picograms per milliliter (pg/mL)
  Day 1: Pre-dose: number analyzed (Participants) | 89 | 44
  Day 1: Pre-dose | 0.00 (0.00) | 0.18 (1.17)
  Day 1: Post-dose: number analyzed (Participants) | 87 | 44
  Day 1: Post-dose | 2.57 (2.35) | 5.64 (4.27)
  Day 14: Pre-dose: number analyzed (Participants) | 86 | 43
  Day 14: Pre-dose | 1.63 (3.06) | 2.77 (4.77)
  Day 14: Post-dose: number analyzed (Participants) | 81 | 42
  Day 14: Post-dose | 5.81 (5.44) | 11.0 (9.74)
  Day 28: Pre-dose: number analyzed (Participants) | 86 | 45
  Day 28: Pre-dose | 2.68 (4.75) | 3.67 (5.59)
  Day 28: Post-dose: number analyzed (Participants) | 82 | 43
  Day 28: Post-dose | 6.41 (6.92) | 10.9 (9.48)

4. Secondary Outcome: Urine Concentrations of VX-371
Time Frame: as for outcome 3
Population: The PK analysis set included all participants who received at least 1 dose of VX-371. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified time points.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | VX-371 + Hypertonic Saline | VX-371 + Placebo
Number analyzed (Participants) | 88 | 45
pg/mL
  Day 1: Pre-dose | 0.0745 (0.699) | 0.00 (0.00)
  Day 1: Post-dose | 7.78 (11.8) | 22.1 (38.4)
  Day 14: Pre-dose: number analyzed (Participants) | 85 | 43
  Day 14: Pre-dose | 41.0 (97.2) | 69.6 (107)
  Day 14: Post-dose: number analyzed (Participants) | 83 | 42
  Day 14: Post-dose | 38.9 (64.8) | 75.0 (98.7)
  Day 28: Pre-dose: number analyzed (Participants) | 84 | 45
  Day 28: Pre-dose | 65.3 (155) | 98.6 (175)
  Day 28: Post-dose: number analyzed (Participants) | 82 | 43
  Day 28: Post-dose | 49.1 (120) | 75.1 (108)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days post last administration of study drug, up to 112 days
Description: Safety set included all participants who received at least 1 dose of inhaled study drug.
Arm/Group | VX-371 + Hypertonic Saline | Hypertonic Saline | VX-371 + Placebo | Placebo
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90 | 0/46 | 0/42
Serious Adverse Events (participants affected / at risk) | 8/89 | 4/90 | 6/46 | 3/42
Other Adverse Events (participants affected / at risk) | 49/89 | 55/90 | 26/46 | 20/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VX-371 + Hypertonic Saline (N=89) | Hypertonic Saline (N=90) | VX-371 + Placebo (N=46) | Placebo (N=42)
Infective pulmonary exacerbation of cystic (Infections and infestations) | 3 | 3 | 5 | 3
Cystic fibrosis related diabetes (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Cystic fibrosis respiratory infection (Surgical and medical procedures) | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VX-371 + Hypertonic Saline (N=89) | Hypertonic Saline (N=90) | VX-371 + Placebo (N=46) | Placebo (N=42)
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 13 | 13 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 4 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 2 | 1
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 3 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 5 | 5
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 5 | 2
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 8 | 12 | 6 | 3
Nasopharyngitis (Infections and infestations) | 0 | 5 | 2 | 2
Alanine aminotransferase increased (Investigations) | 3 | 5 | 0 | 4
Pulmonary function test decreased (Investigations) | 0 | 0 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 3 | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 6 | 1 | 0
Headache (Nervous system disorders) | 6 | 8 | 2 | 1
Pyrexia (General disorders) | 1 | 5 | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-07-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT02709109/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT02709109/SAP_001.pdf